CLINICAL TRIAL: NCT05165992
Title: Nebulized Fentanyl for Respiratory Symptoms in Patients With COVID-19 (Ventanyl Trial)
Brief Title: Nebulized Fentanyl for Respiratory Symptoms in Patients With COVID-19
Acronym: Ventanyl
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MRC-01-21-798
Record Dates: First submitted 2021-12-20; First posted 2021-12-21 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2021-12

CONDITIONS: COVID-19 Pneumonia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Nebulized Fentanyl (Active Comparator): Intervention group (n=100): Administration of nebulized Fentanyl (25 μg in 5 ml of normal saline) over 15 mins, thrice daily using a traditional nebulizer. Treatment duration - 48 hours
  Interventions: Drug: Nebulized Fentanyl
- Nebulized 0.9% Saline Solution (Placebo Comparator): Control group (n=100): Administration of nebulized 0.9% saline solution (5 ml of normal saline), over 15 minutes, thrice daily using a traditional nebulizer. Treatment duration - 48 hours
  Interventions: Drug: Nebulized Fentanyl

INTERVENTIONS:
Drug: Nebulized Fentanyl — Administration of nebulized Fentanyl (25 μg in 5 ml of normal saline) over 15 mins, thrice daily using a traditional nebulizer. Treatment duration - 48 hours

SUMMARY:
Patients with Coronavirus Disease (COVID-19) experience distressing and challenging to manage respiratory symptoms. Interventions such as Oxygen (O2) therapy, oral opiates, and traditional nebulizers like ipratropium bromide and salbutamol, are variably effective, and therapeutic responses in individual patients are difficult to predict. The purpose of this study is to investigate the efficacy of nebulized fentanyl citrate on dyspnea, cough, and throat pain in patients with COVID-19, as well as evaluate the safety with any potential adverse events.

In COVID-19, about 59% of patients will exhibit cough, 35% generalized body ache and sore throat and 31% will have dyspnea. Nebulized Lidocaine, magnesium, and opioids are alternative methods for the management of respiratory symptoms in various patients. Fentanyl nebulization was found to be effective in decreasing dyspnea in chronic obstructive pulmonary disease (COPD) patients by decreasing the rate of spontaneous respiratory rate, modulating cortical activity, and diminishing the brain stem chemoreceptor response to hypoxia and hypercarbia. The investigators hypothesize that nebulized fentanyl is superior to nebulized saline in suppressing cough, respiratory drive, improving breathlessness or dyspnea with the additional advantage of throat pain relief with minimal adverse effects in patients with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 - 65 years
* Confirmed diagnosis (COVID-19) - positive PCR
* Tachypnoea (Respiratory rate> 30/min)
* Ability to provide informed consent and perform all study procedures

Exclusion Criteria:

* History of allergy or adverse reaction to fentanyl or other opioids
* Pregnancy
* Active neuromuscular or musculoskeletal disease.
* Active malignancy
* Morbid obesity (Body mass index >40)
* Use of opioids in the previous 4 weeks.
* Inability to provide informed consent and perform all study procedures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-02 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Breathlessness | 15-minutes post-treatment
  The severity of breathlessness will be measured by the 10-point Borg Scale. Patients will be instructed to use this scale to rate the difficulty of breathing. It starts at number 0 where breathing is causing no difficulty at all and progresses through to number 10 where breathing difficulty is maximal.
Throat Pain | 15-minutes post-treatment
  Throat pain will be graded by the Numerical Rating Scale (NRS), in which patients will be asked to circle the number between 0 and 10, that fits best to their pain intensity. Zero usually represents 'no pain at all' whereas the upper limit represents 'the worst pain ever possible'.
Cough | 15-minutes post-treatment
  The cough severity score represents a simple instrument, using a 10 point scale, where the patient can indicate the severity of their cough between the two extremes: one for no cough while 100 mm is the most severe cough.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad Y Khatib, MD, Principal Investigator — Hamad Medical Corporation

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hildreth L, Pett D, Higgins E. Nebulized fentanyl for refractory dyspnea secondary to chronic obstructive pulmonary disease (COPD): A case report. Respir Med Case Rep. 2020 Oct 12;31:101251. doi: 10.1016/j.rmcr.2020.101251. eCollection 2020. PMID 33145156
- [Background] Foral PA, Malesker MA, Huerta G, Hilleman DE. Nebulized opioids use in COPD. Chest. 2004 Feb;125(2):691-4. doi: 10.1378/chest.125.2.691. PMID 14769753
- [Background] Afolabi TM, Nahata MC, Pai V. Nebulized opioids for the palliation of dyspnea in terminally ill patients. Am J Health Syst Pharm. 2017 Jul 15;74(14):1053-1061. doi: 10.2146/ajhp150893. PMID 28687551
- [Background] Krajnik M, Jassem E, Sobanski P. Opioid receptor bronchial tree: current science. Curr Opin Support Palliat Care. 2014 Sep;8(3):191-9. doi: 10.1097/SPC.0000000000000072. PMID 25010531
- [Background] Boyden JY, Connor SR, Otolorin L, Nathan SD, Fine PG, Davis MS, Muir JC. Nebulized medications for the treatment of dyspnea: a literature review. J Aerosol Med Pulm Drug Deliv. 2015 Feb;28(1):1-19. doi: 10.1089/jamp.2014.1136. Epub 2014 Jun 10. PMID 24914770
- [Background] Benyamin R, Trescot AM, Datta S, Buenaventura R, Adlaka R, Sehgal N, Glaser SE, Vallejo R. Opioid complications and side effects. Pain Physician. 2008 Mar;11(2 Suppl):S105-20. PMID 18443635
- [Background] Uronis HE, Currow DC, Abernethy AP. Palliative management of refractory dyspnea in COPD. Int J Chron Obstruct Pulmon Dis. 2006;1(3):289-304. doi: 10.2147/copd.2006.1.3.289. PMID 18046866
- [Background] Elliott J, Whitaker M, Bodinier B, Eales O, Riley S, Ward H, Cooke G, Darzi A, Chadeau-Hyam M, Elliott P. Predictive symptoms for COVID-19 in the community: REACT-1 study of over 1 million people. PLoS Med. 2021 Sep 28;18(9):e1003777. doi: 10.1371/journal.pmed.1003777. eCollection 2021 Sep. PMID 34582457
- [Background] Scialo F, Daniele A, Amato F, Pastore L, Matera MG, Cazzola M, Castaldo G, Bianco A. ACE2: The Major Cell Entry Receptor for SARS-CoV-2. Lung. 2020 Dec;198(6):867-877. doi: 10.1007/s00408-020-00408-4. Epub 2020 Nov 10. PMID 33170317